CLINICAL TRIAL: NCT06836869
Title: A Multicenter, Non-inferiority Trial to Compare the Effectiveness and Safety of Laparoscopic Radical Hysterectomy Incorporating Modified Tumor-free Techniques Versus Abdominal Radical Hysterectomy in Patients With Stage IB2 Cervical Cancer
Brief Title: Modified Tumor-free Techniques Operation to Cervical Cancer
Acronym: MOTTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Second Hospital of Jilin University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Cangzhou Central Hospital (Other); Zhejiang Cancer Hospital (Other); Hunan Provincial Maternal and Child Health Care Hospital (Other); LanZhou University (Other); RenJi Hospital (Other); The Fourth Military Medical University, Xijing Hospital (Unknown); Affiliated Hospital of Shanxi University of Traditional Chinese Medicine (Unknown); Afﬁliated Hospital of North Sichuan Medical College (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other)
Responsible Party: Principal Investigator, xiang yang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOTTO
Record Dates: First submitted 2025-02-11; First posted 2025-02-20 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-02

CONDITIONS: Cervical Cancer Stage IB2
Keywords: radical hysterectomy; Modified Tumor-Free Techniques; cervical cancer; FIGO stage 1B2; laparotomy; laparoscopic surgery
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center, open-label, blind endpoint evaluation (PROBE), non-inferiority, randomized controlled trial with a parallel-group design. The main hypothesis of this study is that laparoscopic radical hysterectomy incorporating modified tumor-free techniques (LRH-MTF) is non-inferior to abdominal radical hysterectomy (ARH) in terms of disease-free survival at 4.5 years post-operation. A non-inferiority margin of 7% is set based on previous studies. This means that as long as the difference in the 4.5-year disease-free survival rate between LRH-MTF and ARH is within this non-inferiority margin, LRH-MTF will be considered non-inferior to ARH. If LRH-MTF meets this criterion, it can potentially offer the advantages of minimally invasive surgery, such as reduced surgical trauma, shorter hospital stay, and faster recovery, while maintaining comparable oncological outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LRH-MTF (Experimental): Laparoscopic radical hysterectomy incorporating modified tumor-free techniques
  Interventions: Procedure: Laparoscopic radical hysterectomy incorporating modified tumor-free techniques
- ARH (Active Comparator): Abdominal radical hysterectomy
  Interventions: Procedure: Abdominal radical hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic radical hysterectomy incorporating modified tumor-free techniques — Thoroughly examine the pelvic and abdominal cavities. Coagulation of the fallopian tubes are recommanded at the beginning of the surgery. The use of uterine manipulator is prohibited. An "8"-suture at the uterine fundus is recommended. Insert a trocar 3 cm above the pubic symphysis and suspend the uterus by pulling with a needle holder. Alternative methods are also acceptable. Perform pelvic lymphadenectomy. Conduct radical hysterectomy according to the Q-M classification type C. Before incising the vagina, the upper part of the vagina must be closed (using a cable tie or suture), or the vagina can be incised transvaginally after deflating the pneumoperitoneum. Sterilized distilled water or saline solution (≥1000 mL) is used to irrigate the pelvic cavity. The vaginal stump can be sutured either laparoscopically or transvaginally.
  Arms: LRH-MTF
Procedure: Abdominal radical hysterectomy — At the onset of surgery, comprehensively explore the pelvic and abdominal cavities. If intraperitoneal metastases are identified, radical hysterectomy should be aborted. Perform pelvic lymphadenectomy. After lymph node resection, remove the lymph nodes from the surgical field promptly. Sentinel lymph node mapping and biopsy are not performed in this study. Perform radical hysterectomy according to type C of the Q-M classification. It can be accompanied by or without bilateral salpingo - oophorectomy. For patients who retain their ovaries, bilateral ovarian transposition can be carried out. Before incising the vagina, close the upper segment of the vagina and/or the vaginal stump. This can be achieved using instruments such as a large right - angle clamp or an auricular clamp. Sterilized distilled water or saline solution (≥1000 mL) is used to irrigate the pelvic cavity.
  Arms: ARH

SUMMARY:
The goal of this clinical trial is to learn if laparoscopic radical hysterectomy incorporating modified tumor-free techniques (LRH-MTF) works to treat FIGO stage IB2 cervical cancer as good as abdominal radical hysterectomy (ARH). It will also learn about the safety of LRH-MTF. The main questions it aims to answer are:

Does LRH-MTF achieve a non-inferior disease-free survival rate at 4.5 years post - operation compared to ARH? What complications do patients have during and after the operation when receiving LRH-MTF? Researchers will compare LRH-MTF to ARH to see if LRH-MTF works no worse than ARH in treating FIGO stage IB2 cervical cancer.

Participants will:

1. Undergo either LRH-MTF or ARH as assigned by randomization.
2. Visit the hospital for follow-up according to the study schedule for various examinations including blood tests, imaging studies, and assessment of complications.
3. Complete quality-of-life questionnaires such as EORTC QLQ-C30, QLQ-CX24, FSFI, and FSDS-R at baseline (pre-operation) and specific time points during the follow - up period (post-operation 6 months, 1 year, 2 years, 3 years, 4.5 years).

DETAILED DESCRIPTION:
A progress report will be conducted within 4 weeks after all participants have completed their 6-month postoperative visit (the 5th visit). The report will be performed by an independent third-party statistical team, which will provide a comprehensive analysis of the safety data, baseline characteristic, and perioperative indicators.

The study will perform one final analysis.

ELIGIBILITY:
1. Inclusion Criteria:

   1.1 Females aged 18 to 65 years old. 1.2 Histologically confirmed primary cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma.

   1.3 FIGO 2018 stage IB2. 1.4 The maximum diameter of the cervical lesion measured by MRI is >2 cm and ≤4 cm. For those with MRI contraindications, PET/CT, CT, or ultrasound can be used as alternatives.

   1.5 Scheduled to receive type C (Q - M classification) radical hysterectomy. 1.6 Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

   1.7 Willing to participate in this trial and sign the informed consent form. 1.8 Able to cooperate and complete follow - up and relevant examinations. 1.9 For pre - menopausal women, a negative pregnancy test within 30 days before surgery.

   1.10 Laboratory test indicators of vital organs meet the standards
2. Exclusion Criteria:

2.1 Special pathological types (gastric - type adenocarcinoma, neuroendocrine carcinoma, clear cell carcinoma, carcinosarcoma, etc.).

2.2 Imaging examinations suggest pelvic or para - aortic lymph node metastasis (MRI or CT shows a short - axis diameter of ≥1.5 cm, or SUV ≥2.5), or histopathology indicates lymph node metastasis.

2.3 History of pelvic and abdominal radiotherapy. 2.4 History of neoadjuvant chemotherapy. 2.5 Uterus larger than that at 10 weeks of pregnancy. 2.6 Contraindications for surgery and anesthesia (such as severe medical comorbidities).

2.7 Patients who cannot tolerate the Trendelenburg position. 2.8 Patients who cannot cooperate with treatment and follow - up. 2.9 Pregnant patients. 2.10 History of other malignancies, except for those who have been cancer - free for more than 3 years with no current evidence of tumor recurrence.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
4.5-year Disease-free Survival | From enrollment to the 4.5 years after the end of treatment
  The time from randomization until the first recurrence or death from any cause within 4.5 years after surgery. Recurrence needs to be confirmed by histopathology and/or imaging. If pathological evidence cannot be obtained, recurrence should be determined by two or more detection methods, and adjudicated by an independent Endpoint Event Evaluation Committee.

SECONDARY OUTCOMES:
4.5-year Overall Survival | From enrollment to the 4.5 years after the end of treatment
  The time interval from randomization to death from any cause within 4.5 years after surgery.
Pattern of Reccurence | From surgery to the 4.5 years after the end of treatment
  According to the location of the first recurrence, it is divided into intra-pelvic recurrence and distant recurrence. Analyze the differences in the location of tumor recurrence after different surgical methods to provide a reference for subsequent treatment and prognosis judgment.
Estimated surgical blood loss | From the start to the end of the surgery up to 24 hours
  Calculate it as the difference in the weight of gauze/gauze pads before and after the surgery (g) divided by 1.05, plus the difference between the total volume of aspirated fluid and the volume of irrigation fluid at the end of the surgery (mL). Also, record whether blood transfusion is performed during the surgery and within 1 week after the surgery. In addition, record the changes in hemoglobin before and after the surgery to assess blood loss. Perform a complete blood count (hemoglobin) test within 1 week before the surgery and on the 1st day after the surgery.
Operating time | From the start to the end of the surgery up to 24 hours
  The time from making the first incision to completing the suturing.
Postoperative pain | From surgery to the third day after surgery
  It is evaluated using the Visual Analogue Scale (VAS). Additionally, the types, quantities, and administration methods of postoperative analgesics are recorded.
Gastrointestinal function recovery | From the end of surgery to the first postoperative flatus at 7 days.
  Record the time (in hours) of the first postoperative flatus.
Length of hospital stay | From hospitalization to discharge up to 90 days.
  The number of days from hospitalization to discharge.
Treatment cost | From enrollment to the 4.5 years after the end of treatment
  The total cost of hospitalization and outpatient services related to this disease. Conduct cost - effectiveness analysis through incremental cost, improvement of functional outcomes, and quality - adjusted life - years.
EORTC QLQ - C30 scale | From enrollment to the 4.5 years after the end of treatment
  EORTC QLQ - C30 is short for European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30. Each of the 15 subscales of the EORTC QLQ - C30 is scored from 0 to 100.
  For the functional scales (physical, role, emotional, cognitive, and social functioning), higher scores indicate better functioning and thus a better outcome. For the symptom scales (fatigue, nausea and vomiting, pain, etc.) and the global health status/QOL scale, a higher score on the symptom scales means more severe symptoms (a worse outcome), while a higher score on the global health status/QOL scale means a better quality of life. It is used to evaluate the quality of life at baseline (pre - operation) and at 6 months, 1 year, 2 years, 3 years and 4.5 years after surgery.
EORTC QLQ - CX24 Scale | From enrollment to the 4.5 years after the end of treatment
  EORTC QLQ - CX24 Scale is short for European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Cervical Cancer Module. Similar to the QLQ - C30, most of its subscales are scored from 0 to 100. Interpretation of Scores: The interpretation is generally in line with the QLQ - C30. Higher scores in functional aspects indicate better conditions, while higher scores in symptom-related aspects indicate more severe symptoms or worse outcomes. It is used to evaluate the quality of life at baseline (pre - operation) and at 6 months, 1 year, 2 years, 3 years and 4.5 years after surgery.
FSFI Scale | From enrollment to the 4.5 years after the end of treatment
  FSFI is short for Female Sexual Function Index. Minimum and Maximum Values: The total score of the FSFI ranges from 2 to 36. Interpretation of Scores: A higher score indicates better female sexual function and a better outcome in terms of sexual health. Scores below a certain threshold may indicate sexual dysfunction.
  It is used to evaluate the sexual function at baseline (pre - operation) and at 6 months, 1 year, 2 years, 3 years and 4.5 years after surgery.
FSDS - R Scale | From enrollment to the 4.5 years after the end of treatment
  FSDS - R Scale is short for Female Sexual Distress Scale - Revised. Minimum and Maximum Values: The FSDS - R typically has a score range from 0 to 52.
  Interpretation of Scores: In this scale, a higher score indicates a higher level of sexual distress, meaning a worse outcome. It reflects the degree of distress a woman experiences related to her sexual function or situation.
  It is used to evaluate the sexual function at baseline (pre - operation) and at 6 months, 1 year, 2 years, 3 years and 4.5 years after surgery.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hunan Provincial Maternal and Child Health Care Hospital, Changsha, Hunan
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Renji Hospital Affiliated to The Shanghai Jiao Tong University Medical School, Shanghai, Shanghai Municipality
  - Affiliated Hospital of Shanxi University of Traditional Chinese Medicine, Xianyang, Shanxi
  - The Fourth Military Medical University, Xijing Hospital, Xi’an, Shanxi
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Zhejiang cancer hospital, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing
  - Tianjin Central Hospital of Gynecology Obstetrics, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the primary outcome results are published.
Access Criteria: Qualified gynecologists can obtain an IPD by contacting the central contact person.

REFERENCES:
- [Background] Kanao H, Aoki Y, Fusegi A, Omi M, Nomura H, Tanigawa T, Okamoto S, Kurita T, Netsu S, Omatsu K, Yunokawa M. Feasibility and Outcomes of "No-Look No-Touch" Laparoscopic Radical Trachelectomy for Early-Stage Cervical Cancer. J Clin Med. 2021 Sep 15;10(18):4154. doi: 10.3390/jcm10184154. PMID 34575265
- [Background] Chiva L, Zanagnolo V, Querleu D, Martin-Calvo N, Arevalo-Serrano J, Capilna ME, Fagotti A, Kucukmetin A, Mom C, Chakalova G, Aliyev S, Malzoni M, Narducci F, Arencibia O, Raspagliesi F, Toptas T, Cibula D, Kaidarova D, Meydanli MM, Tavares M, Golub D, Perrone AM, Poka R, Tsolakidis D, Vujic G, Jedryka MA, Zusterzeel PLM, Beltman JJ, Goffin F, Haidopoulos D, Haller H, Jach R, Yezhova I, Berlev I, Bernardino M, Bharathan R, Lanner M, Maenpaa MM, Sukhin V, Feron JG, Fruscio R, Kukk K, Ponce J, Minguez JA, Vazquez-Vicente D, Castellanos T, Chacon E, Alcazar JL; SUCCOR study Group. SUCCOR study: an international European cohort observational study comparing minimally invasive surgery versus open abdominal radical hysterectomy in patients with stage IB1 cervical cancer. Int J Gynecol Cancer. 2020 Sep;30(9):1269-1277. doi: 10.1136/ijgc-2020-001506. Epub 2020 Aug 11. PMID 32788262
- [Background] Ramirez PT, Frumovitz M, Pareja R, Lopez A, Vieira M, Ribeiro R, Buda A, Yan X, Shuzhong Y, Chetty N, Isla D, Tamura M, Zhu T, Robledo KP, Gebski V, Asher R, Behan V, Nicklin JL, Coleman RL, Obermair A. Minimally Invasive versus Abdominal Radical Hysterectomy for Cervical Cancer. N Engl J Med. 2018 Nov 15;379(20):1895-1904. doi: 10.1056/NEJMoa1806395. Epub 2018 Oct 31. PMID 30380365
- [Background] Li Y, Zhao J, Ding X, Liang C, Wang W, Ren T, Jiang F, Yang J, Xiang Y. Oncologic Outcomes of Laparoscopic Radical Hysterectomy Incorporating Modified Tumor-Free Techniques. Obstet Gynecol. 2025 Feb 1;145(2):134-143. doi: 10.1097/AOG.0000000000005805. Epub 2024 Dec 19. PMID 39700500